CLINICAL TRIAL: NCT06758427
Title: Hierarchy of Effects of Laboratory Markers and Their Interaction With Comorbidity Concerning Outcome and Personalized Treatment of Trauma Patients in Emergency Care and Rehabilitation
Acronym: HELICOPTER
Status: Not yet recruiting | Type: Observational
Sponsor: Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen, BG Klinik Tu (Other)
Collaborators: BG Klinik Murnau (Unknown); BG Trauma Center Ludwigshafen (Other); BG Klinikum Duisburg (Unknown); BG Klink Hamburg (Unknown); Unfallkrankenhaus Berlin (Other); BG Ambulanz Bremen (Unknown); Bundeswehrkrankenhaus Ulm (Unknown); Paracelsus Universität Salzburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: HELICOPTER
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Complications; Surgical Site Infection; Wound Infection; Non-healing Wound; Pseudarthrosis; Bone Infection; Pneumonia; Nosocomial Infection
Keywords: long bone fracture, trauma
MeSH Terms: conditions — Postoperative Complications; Surgical Wound Infection; Wound Infection; Pseudarthrosis; Pneumonia; Cross Infection; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At least ten percent of trauma patients suffer from any sort of complication. The study aims to identify a risk factor profile to early identify trauma patients at risk.

DETAILED DESCRIPTION:
Trauma patients suffer from a high risk of complications that ranges from soft tissue complications, surgical site infection till bone non-union. Comorbidities are often know to be associated with complications. Also certain blood markers could be identified to be an indicator.

However, certain risk factors have only been investigated in small trauma cohorts so far. This study is a prospective multi center cohort trail that aims to collect all clinical data, comorbidities, medication, blood markers in trauma patients after long bone fractures. In a 6 months and one year follow up patients with complications will be identified. Methods of machine learning will help to identify a risk factor profile for certain groups of patients with complications.

The aim of the study is to early identify patients at risk for a complication after trauma according to their blood marker, clinical, comorbidity and medication profile.

ELIGIBILITY:
Inclusion Criteria:

* acute long bone fracture (humerus, ulna, radius, femur, tibia) with surgical treatment

Exclusion Criteria:

* associated severe injury (ISS > 16)
* associated traumatic brain injury
* associated traumatic spine injury
* dementia

Ages: 18 Years to 67 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients that suffer from an acute lone bone fracture, require surgical treatment and belong to the age group of being able to working (18 - 67 years old)
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
any complication after long bone fracture | 6 months, one year
  number of patients that suffer from a complication after surgical treatment of a primary long bone fracture
Clavien Dindo Classification | 6 months, one year
  Clavien Dindo Classification classifies surgical complications. All patients will be classified according to Clavien Dindo after 6 months and one year.

SECONDARY OUTCOMES:
Charlson Comorbidity Index (CCI) | Initially
  Charlson Comorbidity Index classifies comorbidities of patients. All particiapants will be screened for their comorbidities and classified according to CCI.
number of medications | initally
  Intake of medication will be assessed and number of medication will be identified.
EuroQual 5 Dimensions Questionnaire (EQ5D5L) | initially, 6 months, one year.
  EQ5D5L will be assessed from each participant to identify their quality of life.
patient reported outcome measure associated with the lone bone fracture | initially, 6 months, one year.
  patient reported outcome measure will be assessed by each patient that is associated with the lone bone fracture

CONTACTS AND LOCATIONS:
Overall Officials: Marie K Reumann, MD, Principal Investigator — Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen
Locations (1):
- Department of Trauma and Reconstructive Surgery at Eberhard Karls University Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Data of all patients will be pseudonymised. No individual participant data will be identified.